CLINICAL TRIAL: NCT05798039
Title: Colorado Nurse Family Heart Trial for the ENRICH Program
Brief Title: ENRICH Nurse-Family Partnership Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-0021; UG3HL162967 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Blood Pressure; Body Composition; Blood Sugar; Body Weight; Diet Habit; Physical Inactivity
MeSH Terms: conditions — Body Weight; Feeding Behavior; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENRICHed NFP (Experimental): Participants will receive additional heart health-focused materials and guidance in sessions with their nurse home visitor. The nurse will help them choose and work towards behavior goals to support their health. This will include goals for activity, diet, weight, blood pressure, diabetes, smoking, social relationships, sleep, parenting, and getting health care.
  Interventions: Behavioral: ENRICH

INTERVENTIONS:
Behavioral: ENRICH — Participants will receive additional heart health-focused materials and guidance in sessions with their nurse home visitor. The nurse will help them choose and work towards behavior goals to support their health. This will include goals for activity, diet, weight, blood pressure, diabetes, smoking, social relationships, sleep, parenting, and getting health care.
  Other Names: NFP-Heart

SUMMARY:
The overarching goal of the proposed study is to develop and test an enrichment to Nurse-Family Partnership (NFP) using an existing, evidence-based program to improve clients' and their children's cardiovascular health from early pregnancy to 24 months postpartum. With support from NFP supervisors and nurses, the investigators will develop new NFP materials promoting healthy diet, activity, sleep, and smoking behaviors, along with optimal weight, glycemia, lipid, and blood pressure profiles. The investigators will conduct a pilot study with up to 40 NFP clients (or women similar to NFP client population) and their nurses to determine feasibility and acceptability of the materials and study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or <24 months postpartum
* Aged 18 years or older
* English- or Spanish-speaking

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Maternal BMI | Enrollment
  Height and weight will be measured and combined to report BMI

SECONDARY OUTCOMES:
A1C | Enrollment
  Blood draw
Blood pressure | Enrollment
  automatic blood pressure monitor will be used to measure both systolic and diastolic blood pressure
Diet Quality | Enrollment
  Diet will be assessed with 24-hour dietary recalls using the Automated Self-Administered system (ASA24). This system uses the USDA multiple-pass method to query all foods and supplements consumed in the prior 24 hours and produces daily and individual food estimates for macronutrients, micronutrients, and MyPyramid Equivalents (such as servings of vegetables, fruits, whole grains, solid fats, and added sugars)
Physical Activity | Enrollment
  Assessed using the Pregnancy Physical Activity Questionnaire (PPAQ), while adjusting metabolic task equivalents for pregnancy. Investigators will calculate average activity intensity (sedentary to vigorous) and type (household, occupational, exercise, transportation) over the past 3 months at collection point. Physical activity outcomes include daily minutes of sedentary, light, moderate, vigorous, household, occupational, exercise, transportation activity.
Smoking frequency | Enrollment
  Participants will be asked about lifetime and recent (past 6 months) usage of cigarette and marijuana. Smoking outcomes include any smoking in pregnancy (binary) and number of cigarettes (total, trimester-specific).
Maternal adiposity | Enrollment
  Percent of total mass that is fat mass, as measured by air displacement plethysmography using the BOD POD device
Sleep Quality | Enrollment
  Assessed using a sleep questionnaire developed and validated by the NIH Patient Report Outcome Information System (PROMIS), adapted for this study. This form queries daytime and nighttime sleep start times, stop times, and duration, and also collect data on sleep disturbances and sleep-related impairments (trouble falling asleep, staying asleep, number of nighttime awakenings, feeling refreshed upon waking, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Allison, MD, MSPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No